CLINICAL TRIAL: NCT01625143
Title: Molecular Taxonomy of Pediatric Cancer
Brief Title: Studying Genes in Samples From Younger Patients With Relapsed Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AALL12B7; NCI-2012-01976 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000735342 (Other: Clinical Trials.gov); COG-AALL12B7 (Other: Children's Oncology Group)
Record Dates: First submitted 2012-06-17; First posted 2012-06-21 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: B-cell Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia; Untreated Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Archived bone marrow samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: Archived bone marrow samples, collected at the time of diagnosis and relapse, are analyzed for gene expression and histone modifications by microarray, chromatin immunoprecipitation (ChIP) sequencing, and quantitative real-time polymerase chain reaction (qRT-PCR).
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This laboratory study is looking into genes in samples from younger patients with relapsed acute lymphoblastic leukemia. Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors find better ways to treat cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To identify global changes in the epigenome and various underlying histone modifications that characterize relapsed acute lymphoblastic leukemia (ALL).

II. To identify specific transcription factor-binding sites associated with histone alterations.

III. To correlate gene expression changes of differentially regulated genes at relapse with underlying chromatin modifications.

OUTLINE:

Archived bone marrow samples, collected at the time of diagnosis and relapse, are analyzed for gene expression and histone modifications by microarray, chromatin immunoprecipitation (ChIP) sequencing, and quantitative real-time polymerase chain reaction (qRT-PCR).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of B-cell acute lymphoblastic leukemia

  * Paired diagnosis-relapse primary patient samples obtained from the Children's Oncology Group (COG) cell bank

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Diagnosis of B-cell acute lymphoblastic leukemia
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Cellular origins of relapse and the underlying epigenetic mechanisms associated with drug resistance | 1 month
Genes associated with histone modification | 1 month
Biological pathways involved in relapse | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: William Carroll, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States